CLINICAL TRIAL: NCT05107271
Title: Comprehensive Assessment of Intermediate and Long-term Sequelae of COVID-19 Infection and Immunological Correlates of Protection Induced by COVID-19 Vaccines in Patients With Liver Disease: A Prospective Cohort Study.
Brief Title: Evaluation of Long Haul COVID-19 and Vaccine Immunogenicity in Patients With Liver Disease
Acronym: EvaLongCovid
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: 2021-5859
Record Dates: First submitted 2021-11-03; First posted 2021-11-04 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: COVID-19; Chronic Liver Failure; Cirrhosis, Liver; Portal Hypertension; Liver Transplant Disorder
MeSH Terms: conditions — COVID-19; End Stage Liver Disease; Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples will be assessed for serosurvey
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Chronic Liver Disease
  Interventions: Diagnostic Test: COVID-19 serosurvey
- Post Liver Transplantation
  Interventions: Diagnostic Test: COVID-19 serosurvey

INTERVENTIONS:
Diagnostic Test: COVID-19 serosurvey — COVID-19 related antibody testing to assess immunogenicity of COVID-19 vaccines or post natural infection acquired immunity

SUMMARY:
The project is essential to understand the impact of the COVID-19 pandemic in patients with Chronic Liver Disease (CLD).

The impact has been felt due to direct risk of COVID infection in self, or in caregivers, lack of access to services during lockdown, interruptions in transplant listing and waitlist mortality. Briefly, the following points will be focused during the study.

1. Long haul COVID-19 related symptoms.
2. Impact on health and delay in interventions or drug therapy due to interruption of physical outpatient services.
3. Impact on emergency admissions due to refractory ascites, new decompensation, variceal bleeding etc
4. Impact on delayed transplant listing and waitlist mortality
5. Impact on post-transplant patients with lack of access to drug monitoring/ physical OPD
6. Impact on delay in interventions due to hepatobiliary malignancy.
7. Effects of COVID-19 infection, vaccination (single dose, two doses) and no vaccination and protective antibody levels in patients with chronic liver disease and post-transplant recipients.
8. Determination of dose protocol and need for booster vaccination in patients with CLD and post liver transplant recipients.

DETAILED DESCRIPTION:
* The novel coronavirus 2019 (COVID-19) disease, caused by the severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2), has resulted in a devastating global pandemic, with 179,686,071confirmed COVID-19 cases, which include 3,899,172 deaths reported by the World Health Organization1 as of June 25, 2021. As of June 23, 2021, 2,624,733,776 doses of vaccine have been administered globally. COVID-19 has been reported as an air- and surface-borne contagious disease with features of viral pneumonia (fever, cough, lymphopenia, prothrombotic tendency, ground glass opacities on chest radiology) and hypoxemia.
* In addition, alterations in liver chemistries have been reported in patients with and without liver disease, with some reports of increasing severity, complication, and new decompensation, while others refute this possibility. Liver chemistry changes are more likely in those with severe disease and those who have received multiple therapies, requiring high flow oxygen or invasive ventilation.
* Long-term prospective follow-up studies on persistent symptoms, lung function, physical, and psychological problems of discharged patients with cirrhosis, liver failure or liver transplant recipients are urgently required.
* Health care professionals require predictive models of severity of disease and assess the impact of the COVID-19 pandemic on the health of patients with chronic liver disease (CLD), access to care, specialty interventions like endoscopy, and transplantation.
* In addition, the association between liver chemistries, need for invasive ventilation and COVID-19-associated hospital deaths remains controversial and despite availability of breakthrough vaccines, the pandemic is likely to continue claiming more lives.7 Given the heterogenous clinical presentation, the spectrum of liver involvement varies from altered liver chemistry in patients without underlying liver disease to progressive decompensation in patients with cirrhosis.
* Differential access to COVID-19 care may affect outcomes in patients with CLD. Access to care in India may be affected, for example, by age, region of origin, gender, economic status, disability, homelessness, language, digital accessibility, and social factors influencing attitudes to modern medicine. COVID care models deploy multidisciplinary telemedicine clinics to assess physical and mental health symptoms and to conduct appropriate investigations by calling patients for physical consultation, there has been a barrier to access to care and interventions over the course of the COVID-19 pandemic in India.
* Patients have suffered increased waitlist mortality due to reduction in the access to affordable transplant and redistribution of priority resources to the COVID-19 effort. Patients who are liver transplant (LT) recipients have also suffered from lack of access to follow up due to logistic concerns and travel restrictions. The incidence of COVID-19 infection and outcomes in this subgroup is still unknown. This requires data and policy making at the National level based on serosurveys and vaccination success in our CLD population.
* Patients with chronic liver disease who have suffered from COVID-19 need access to rehabilitation services, with an integrated, multidisciplinary service, based on local need and resources. A range of specialists should be available, especially for expertise in treating fatigue and respiratory symptoms (including breathlessness); additional expertise may be sourced depending on the age and symptoms of the person. The incidence of post COVID-19 fungal sepsis in patients of CLD and LT recipients is another point of concern, and data regarding this secondary effect in our patient cohort is still unknown.
* A major gap in delivery of care is the disruption of the seamless referral pathways between primary care and tertiary level centres. Due to the digital divide between urban and rural sectors, the access to routine services like endoscopy, preventive health care checks, rehabilitation services, transplantation services, endoscopy and interventional radiology procedures and mental health care in our patient cohort has been noted but not systematically evaluated.
* Lastly, about 10% of patients with COVID-19 infection may suffer persistent symptoms, and resulted in a large cohort of individuals with long haul COVID symptoms. The effect of COVID-19 on health care systems and society will be noted for years to come, and a systemic study on the burden of the problem needs to be undertaken to formulate appropriate health care policy.

ELIGIBILITY:
Inclusion Criteria:

1. The person is between the ages of 18-75 years at the time of signing the informed consent form.
2. Individual has chronic liver disease of any etiology and is attached to the Hepatology services of the PGIMER, Chandigarh.
3. Individual has had a positive SARS-COV-02 test (PCR) within the last 12 months or has been diagnosed presumptive positive and has been treated for COVID-19 within the last 12 months.
4. Individual has not fully recovered from COVID-19 in weeks or months despite a negative Sars-COV-02 test and has been diagnosed with Post COVID-19 syndrome.
5. Individual is experiencing 2 or more symptoms for over 12 weeks either continually or intermittently with relapses not experienced pre-illness, that interferes with normal daily activities. Symptoms must be new symptoms, or dramatic worsening of symptoms i.e., subject did not have symptoms, and had not sought medical treatment for the symptoms prior to COVID-19, or the symptoms are dramatically worse (in severity and frequency).

   * Extreme fatigue - feeling overtired with low energy and a strong desire to sleep.
   * Shortness of breath - (dyspnea) a feeling of being winded, difficulty in breathing, or a hunger for air.
   * Cough - hacking, or dry barking sound lingering dry or wet.
   * Brain fog -a diminished mental capacity marked by the inability to concentrate or to think or reason clearly that interferes with daily activities.
   * Headache - Sharp or dull reoccurring or intermittent that were not present pre-illness.
   * Body aches - muscle soreness or generalized achiness throughout the body.
   * Joint pain - pain in the joints due to inflammation not experienced before illness.
   * Chest pain - (angina) feeling pressure, fullness, or tightness in your chest
   * Sleep issues - any sleep disturbances in sleep quality that makes sleep see inadequate or unrefreshing like insomnia or hypersomnia.
   * Loss of Taste/Smell - Diminished sense of taste or smell.

Exclusion Criteria:

1. Subject is unable to provide informed consent or to comply with study requirements.
2. Subject has currently been diagnosed with active COVID-19 disease.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Liver Disease or those who are post LT recipients who are attached to the inpatient, outpatient, and telehealth services of the Department of Hepatology, PGIMER Chandigarh will be screened for inclusion
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Long haul COVID-19 related symptoms | 1 year
  'Long-COVID-19' describes the long duration symptoms that patients who have recovered from COVID-19 continue to experience even in their post-recovery phase
Immunogenicity of vaccine | 1 year
  Effects of COVID-19 infection, vaccination (single dose, two doses) and no vaccination and protective antibody levels in patients with chronic liver disease and post-transplant recipients

CONTACTS AND LOCATIONS:
Overall Officials: Virendra Singh, MD DM, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided